CLINICAL TRIAL: NCT05575518
Title: A Pragmatic Trial With Optimized Dose of Rifampicin and Moxifloxacin for the Treatment of Drug Susceptible Pulmonary Tuberculosis
Acronym: OptiRiMoxTB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stellah Mpagama (Other Government)
Collaborators: University of St Andrews (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Stellah Mpagama, Director of Research, Kibong'oto Infectious Diseases Hospital
Organization: Kibong'oto Infectious Diseases Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OptiRiMoxTB-01
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Tuberculosis; Human Immunodeficiency Virus
Keywords: TB/HIV; Phase III; Randomised
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No intervention (No Intervention): Standard of care according to the National TB Programmes which is a weight-banded rifampicin, isoniazid, pyrazinamide, and ethambutol for weeks 0-8 followed by rifampicin and isoniazid for weeks 9-26.
- Experimental Arm 1 (Experimental): Optimised dose of rifampicin. The rifampicin 35mg/kg alongside standard weight-banded doses of isoniazid, pyrazinamide, and ethambutol, once daily
  Interventions: Drug: Optimised rifamycin
- Experimental Arm 2 (Experimental): Optimised dose of rifampicin and moxifloxacin. The rifampicin 35mg/kg and moxifloxacin 400mg alongside standard weight-banded doses of isoniazid and pyrazinamide, once daily.
  Interventions: Drug: Optimised rifamycin

INTERVENTIONS:
Drug: Optimised rifamycin — optimised dose rifampicin with or without moxifloxacin
  Other Names: 8-methoxy-fluoroquinolone
  Arms: Experimental Arm 1; Experimental Arm 2

SUMMARY:
Tuberculosis (TB) remains a major global public health problem, particularly in low- and middle-income countries (LMICs) in Africa, Asia, and Eastern Europe. Approximately 10 million people fall sick with TB, causing up to 2 million deaths, worldwide per year. Considerable progress was made in TB control from 1990-2015, motivating the World Health Organization (WHO) to launch an ambitious EndTB strategy. However, the effect of the ongoing Coronavirus Disease 2019 (Covid-19) pandemic has been devastating and the last two years have seen the first year-on-year increases (of 5.6%) in TB mortality since 2005 . In order to regain lost ground, and re-establish progress towards elimination of TB, innovation is needed in all aspects of TB control, including development of shorter treatment regimens for drug susceptible (DS) and multi-drug resistant / rifampicin resistant (MDR/RR) forms of the disease.

This protocol seeks to conduct the TB clinical trial combining the 8-methoxyfluroquinolone and optimised dose of rifamycing to address two questions. The first is to confirm the non-inferiority of a four-month optimised dose rifamycin and moxifloxacin-based regimen amongst African TB patient populations with high rates of co-incident HIV. Secondly, we seek to establish that the rifamycin of choice in potent 4-month anti-TB treatments could be rifampicin as this will be more rapidly up-scalable for public health impact.

DETAILED DESCRIPTION:
The study objectives of this clinical trial are

Primary effectiveness objective: To evaluate whether one or both of two experimental regimens based on optimised dose rifampicin with or without moxifloxacin and given for 16 weeks are non-inferior to standard treatment for drug-susceptible tuberculosis given for 26 weeks, as assessed by patient survival, free of tuberculosis 12 months after initiation of therapy.

Primary safety objective: To evaluate whether one or both of two experimental regimens based on optimised dose rifampicin with or without moxifloxacin and given for 16 weeks are as safe and tolerable as standard treatment for drug-susceptible tuberculosis given for 26 weeks, as assessed by the frequency of Adverse Events (AEs) of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 severity or higher.

Participants will be individuals with bacteriological confirmed pulmonary TB aged 18 years or above, with or without HIV co-infection in Gabon, Malawi, Mozambique and Tanzania. The trial sites are also established members of the PanACEA / SimpliciTB group including the Centre de Recherches Médicales de Lambaréné (CERMEL)-Gabon, the Helse Nord Tuberculosis Initiative (HNTI) at Kamuzu University of Health Sciences (KUHES)-Malawi and the Polana Caniço Health Research and Training Center (CISPOC) at the Instituto Nacional de Saúde (INS)-Mozambique and the Kibong'oto Infectious Diseases Hospital-Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must meet all the following inclusion criteria prior to enrolment into the trial:

  1. The patient has given fully informed, signed written or witnessed oral informed consent for study participation prior to all trial-related procedures, including HIV testing if HIV status is not known.
  2. The patient has a diagnosis of pulmonary TB established by Xpert MTB/RIF® result which confirms "low" "medium" or "high" level detection of M tuberculosis and does not detect rifampicin resistance.

     1. If the patient has been referred from a clinic at which the pre-screening clinical diagnostic test for TB was an Xpert MTB/RIF® assay done at the trial laboratory, and the full read-out of that result is available, the test does not need to repeated to confirm eligibility.
     2. If the patient has been referred from a clinic at which the pre-screening clinical diagnostic test for TB was an Xpert MTB/RIF® assay done at a non-trial laboratory, but the full read-out of that result is available, the test does not need to repeated to confirm eligibility.
     3. If the patient has been referred to the study from a clinic from which the full pre-screening clinical diagnostic Xpert MTB/RIF® test result is unavailable, a repeat Xpert MTB/RIF® assay should be performed by the study laboratory to confirm eligibility before recruitment.
  3. The patient should be aged ≥ 18 years on the day of providing informed consent.
  4. The patient has a body weight in light clothing and without shoes of at least 35kg.
  5. Female patients of child-bearing potential must have a negative urine or serum pregnancy test ≤ 7 days prior to screening, and consent to practice an effective method of contraception until completion of therapy.
  6. The patient must have a verifiable residence location and telephone number that is accessible if necessary for contact during follow-up.

Exclusion Criteria:

* Patients for whom one of the following criteria is met will be excluded from the trial:

  1. There is concern about any circumstances that raise concern about free, informed consent to study participation.
  2. The patient's pre-screening or screening Xpert MTB/RIF® assay result is "negative","trace", or "very low" positive.
  3. At least one M tuberculosis isolate, either cultured or detected through molecular assays from sputum obtained from the patient prior to treatment initiation is found to be resistant to one or more of: rifampicin, isoniazid, pyrazinamide, ethambutol, or fluoroquinolones (late exclusion).
  4. The patient is in poor general condition where delay in treatment cannot be tolerated, or death within three months is likely, as assessed by the investigator.
  5. The patient had a nose/throat swab which was positive for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV2), on Polymerase Chain Reaction (PCR) or a rapid diagnostic test ≤ 14 days preceding study recruitment.
  6. The patient is pregnant or breast-feeding (female patients only).
  7. The patient is unable to take oral medications.
  8. The patient has received any investigational drug in the past three months.
  9. The patient has received more than five days of treatment directed against active tuberculosis ≤ 6 months preceding initiation of study drugs.
  10. The patient has known intolerance to any of the study drugs, or conditions for which they are contra-indicated.
  11. The patient is unwilling, or unable to adhere to requirements regarding restricted use of other medications during the study. Restricted medications will include medications which prolong the QTc interval, and CYP450 inhibitors or inducers.
  12. The patient is due to initiate, or requires continuation of, non-efavirenz, non-dolutegravir-based anti-retroviral therapy for HIV infection.
  13. The patient has decompensated liver disease and/or aminotransaminases >3x upper limit of normal (ULN), serum total bilirubin level >1.5x ULN or serum/plasma creatinine level >x2 ULN.
  14. The patient has a baseline QTc interval of >450ms.
  15. The patient is being, or about to be, treated for malaria.
  16. The patient has other medical conditions that, in the investigator's judgement, make study participation not in the individual's best interest.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Bacteriological cure, absence of either TB treatment failure or relapse | Participant survival, free of tuberculosis 12 months after randomisation
  Treatment failure, defined as submitting two sputum samples with positive culture for M tuberculosis on different visits, when the first of these samples was collected at or after two weeks prior to the scheduled end of treatment.
  TB relapse, defined as submitting two sputum samples with positive culture for M tuberculosis on different visits, when the first of these samples was collected after completion of scheduled TB therapy and where at least one of the M tuberculosis isolates is genetically similar to the baseline strain.
Proportional of adverse events (AE) of grade 3 severity or higher | 4 or 6 months of treatment
  The severity of all AEs will be classified according to the U.S. National Institutes of Health Common Terminology Criteria for Adverse Events 5.0 (CTCAE).

SECONDARY OUTCOMES:
Proportional of clinically significant adverse events related to the intervention | 4 or 6 months of treatment
  Treatment discontinuation or interruption related to AE
Clinical improvement of TB symptoms | 12 month after randomisation
  Clinical response of TB symptoms as measured by questionnaire
Clinical improvement of body mass index (BMI) | 12 month after randomisation
  Increase of BMI as measured by the ratio of weight (kg) and height squared in metres squared
Clinical improvement of participant reported health status | 12 month after randomisation
  Increase of participant reported health status as measured by questionnaire

OTHER OUTCOMES:
Participant survival free of TB | 12 months after completing TB treatment
  Recurrent of symptoms and bacteriological confirmation of TB

CONTACTS AND LOCATIONS:
Locations (1):
- Kibong'oto Infectious Diseases Hospital, Moshi, Kilimanjaro, Tanzania

REFERENCES:
- [Background] World Health Organization. Global Tuberculosis Report 2021. World Health Organisation 2021.https://www.who.int/publications/i/item/9789240037021
- [Background] World Health Organisation. WHO End TB Strategy: Global strategy and targets for tuberculosis prevention, care and control after 2015. World Health Organization 2021. https://www.who.int/tb/strategy/End_TB_Strategy.pdf
- [Background] Pai M, Kasaeva T, Swaminathan S. Covid-19's Devastating Effect on Tuberculosis Care - A Path to Recovery. N Engl J Med. 2022 Apr 21;386(16):1490-1493. doi: 10.1056/NEJMp2118145. Epub 2022 Jan 5. No abstract available. PMID 34986295
- [Background] Boeree MJ, Diacon AH, Dawson R, Narunsky K, du Bois J, Venter A, Phillips PP, Gillespie SH, McHugh TD, Hoelscher M, Heinrich N, Rehal S, van Soolingen D, van Ingen J, Magis-Escurra C, Burger D, Plemper van Balen G, Aarnoutse RE; PanACEA Consortium. A dose-ranging trial to optimize the dose of rifampin in the treatment of tuberculosis. Am J Respir Crit Care Med. 2015 May 1;191(9):1058-65. doi: 10.1164/rccm.201407-1264OC. PMID 25654354
- [Background] Te Brake LHM, de Jager V, Narunsky K, Vanker N, Svensson EM, Phillips PPJ, Gillespie SH, Heinrich N, Hoelscher M, Dawson R, Diacon AH, Aarnoutse RE, Boeree MJ; PanACEA Consortium. Increased bactericidal activity but dose-limiting intolerability at 50 mg.kg-1 rifampicin. Eur Respir J. 2021 Jul 8;58(1):2000955. doi: 10.1183/13993003.00955-2020. Print 2021 Jul. PMID 33542056
- [Background] Boeree MJ, Heinrich N, Aarnoutse R, Diacon AH, Dawson R, Rehal S, Kibiki GS, Churchyard G, Sanne I, Ntinginya NE, Minja LT, Hunt RD, Charalambous S, Hanekom M, Semvua HH, Mpagama SG, Manyama C, Mtafya B, Reither K, Wallis RS, Venter A, Narunsky K, Mekota A, Henne S, Colbers A, van Balen GP, Gillespie SH, Phillips PPJ, Hoelscher M; PanACEA consortium. High-dose rifampicin, moxifloxacin, and SQ109 for treating tuberculosis: a multi-arm, multi-stage randomised controlled trial. Lancet Infect Dis. 2017 Jan;17(1):39-49. doi: 10.1016/S1473-3099(16)30274-2. Epub 2016 Oct 26. PMID 28100438
- [Background] Dorman SE, Nahid P, Kurbatova EV, Phillips PPJ, Bryant K, Dooley KE, Engle M, Goldberg SV, Phan HTT, Hakim J, Johnson JL, Lourens M, Martinson NA, Muzanyi G, Narunsky K, Nerette S, Nguyen NV, Pham TH, Pierre S, Purfield AE, Samaneka W, Savic RM, Sanne I, Scott NA, Shenje J, Sizemore E, Vernon A, Waja Z, Weiner M, Swindells S, Chaisson RE; AIDS Clinical Trials Group; Tuberculosis Trials Consortium. Four-Month Rifapentine Regimens with or without Moxifloxacin for Tuberculosis. N Engl J Med. 2021 May 6;384(18):1705-1718. doi: 10.1056/NEJMoa2033400. PMID 33951360
- [Background] WHO consolidated guidelines on tuberculosis: Module 4: Treatment - Drug-susceptible tuberculosis treatment [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK581329/ PMID 35727905
- [Derived] Mlyuka HJ, Liyoyo A, Nyaulingo B, Mpolya E, Kaswaga OL, Semvua H, Lwambura S, McHugh TD, Wildner L, Sabiiti W, Adegbite BR, Nliwasa M, Khosa C, Mbelele P, Mbeya B, Jeremiah K, Boeree MJ, Gillespie SH, Sloan DJ, Mpagama SG; SimpliciTB Consortium. A pragmatic trial with an optimized dose of rifampicin and moxifloxacin for the treatment of drug-susceptible pulmonary tuberculosis: a study protocol for open-label, randomized phase III trial (OptiRiMoxTB). Trials. 2026 Jan 30. doi: 10.1186/s13063-026-09466-0. Online ahead of print. PMID 41612490